CLINICAL TRIAL: NCT03322618
Title: Evaluation of the Expression and Functions of the KIR3DL2 Receptor and the Anti-inflammatory Activity of IPH4102 (Monoclonal Antibody IPH4102 Targeting KIR3DL2) in Blood Samples Taken From Patients With Axial Spondyloarthritis and Healthy Volunteers
Brief Title: Evaluation of the Expression and Functions of the KIR3DL2 Receptor and the Anti-inflammatory Activity of IPH4102 in Blood Samples
Acronym: KIR3DL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-33; 2017-A01705-48 (Other: N°IDRCB)
Record Dates: First submitted 2017-10-17; First posted 2017-10-26 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Axial Spondyloarthritis (axSpA); Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SpA HLA-B27 +, (Experimental)
  Interventions: Biological: blood samples
- SpA HLA-B27- (Experimental)
  Interventions: Biological: blood samples
- healthy subject (Active Comparator)
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — 7 tubes of 6 ml (42 ml of blood )

SUMMARY:
the main objectives are

1. to study the pathophysiological role of KIR3DL2 in axSpA and its relationship with Th17 immunity in HLA-B27 + and HLA-B27- patients and
2. to assess the effect on the pro-inflammatory immune response of a cytotoxic monoclonal antibody IPH4102 (anti-KIR3DL2) in these patients.

The study will be carried out on blood samples from 24 patients with axSpA, 12 HLA-B27 + and 12 HLA-B27-, without any drug injection nor direct therapeutic benefit for the participating patients and 12 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of the patient signed before any procedure planned to the protocol
* SPA axial according to the criteria of the ASAS (international Assessment of SpondyloArthritis Society)
* Known Status HLA B27
* Disease activates with a score of BASDAI = 4/10. The BASDAI (Bath Ankylosing Spondylitis Disease Activity Score) is a composite indication(index), validated, used in the therapeutic essays and in current practice for the evaluation of the activity of the SPA.
* Naive Patients of thorough treatment
* Patients of 18 and more years old

Exclusion Criteria:

* Minors
* Pregnant or breast-feeding Women
* Adults under guardianship
* People staying in a sanitary or social establishment
* People in emergency situation
* Not profitable People of a national insurance scheme
* Private persons of freedom
* Treatment by corticoids during the last 30 days before the inclusion
* Treatment by anti-TNF or quite different biomedicine
* Treatment by sulfasalazine
* Reached concomitant by another active chronic inflammatory disease
* Infection chronicles by VHB, VHC or HIV
* Patients included in another study of clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Characterize the present various immunizing populations in patients' blood SPA HLA-B27 + and HLA-B27-(Lymphocytes T CD4 (Th1 Th2, Th17, Tregs), lymphocytes T CD8, cells NK, lymphocytes B, monocytes) | 12 MONTHS
  by flow cytometry.

SECONDARY OUTCOMES:
Expression of the receivers involved in SPA on lymphocytes T CD4 in percentage of cells T CD4 expressing this markers | 12 MONTHS
Dosage of cytokines | 12 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: jean olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France